CLINICAL TRIAL: NCT01100190
Title: A Prospective Study of the NUVANCE Facial Rejuvenation System for Mid-Face, Neck and Jowl Rejuvenation Procedures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in business priorities.
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200-08-001
Record Dates: First submitted 2010-04-07; First posted 2010-04-08 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Ptosis of the Neck, Mid-face and/or Jowl
Keywords: Facelift; Rhytidectomy; Ptosis
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NUVANCE Facial Rejuvenation System (Experimental)
  Interventions: Device: NUVANCE Facial Rejuvenation System

INTERVENTIONS:
Device: NUVANCE Facial Rejuvenation System — The NUVANCE™ Facial Rejuvenation System is a partially absorbable porous mesh device implant with applicator.

SUMMARY:
The objective of this study is to evaluate the clinical tolerability of the NUVANCE™ Facial Rejuvenation System for correcting neck, mid-face and/or jowl ptosis.

DETAILED DESCRIPTION:
This is a multicenter, prospective, single-arm study. The primary tolerability endpoint will be evaluated up to 30-days post-operatively. Secondary endpoints will be evaluated at 6-months. Extended follow-up will be conducted at 12-months, 24-months, and 36-months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject older than 18 years.
* Subject is a candidate for minimally invasive, bilateral facial rejuvenation procedure using NUVANCETM Facial Rejuvenation System according to the device Instructions for Use (IFU).
* Subject is willing and able to provide informed consent and follow study-related requirements.

Exclusion Criteria:

* Subject who previously received surgical facial cosmetic treatment (procedure involving an incision):

  1. Within the last 12 months under the area of the forehead;
  2. Within the last 3 months within the area of the forehead where forehead is defined as the area above the imaginary anatomical line between the lateral canthus of the eye and the upper pole of the ear.
* Subject who previously received a cosmetic procedure with a dermal filler device and/or neurotoxin complex injectable within the last 9 months.
* Subjects with a permanent facial implant.
* Subjects planning on a cosmetic procedure with a permanent implant within 6-months of procedure.
* Subjects planning on a cosmetic procedure with a dermal filler device and/or neurotoxin complex injectable within 6-months of procedure.
* Subjects with significant ptosis where skin excision would be necessary.
* Subject has an active infection (e.g. acne, herpes zoster) or inflammation (e.g. psoriasis, pemphigus vulgaris, cutaneous lupus erythematosus) affecting facial skin.
* Subject has a history of a disorder that can affect wound healing (e.g. subjects pre-disposed to infection or history of keloid formation).
* Subject with pre-existing facial abnormalities (e.g. deformities, Bell's palsy, scarring)
* Subject with a significant psychiatric disorder judged by the clinical investigator that will interfere with the procedure
* Any pre-operative findings that the surgeon identifies that makes the subject not a candidate for a minimally invasive facial cosmetic surgical procedure.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-03-01 (Actual); Primary Completion 2011-04-01 (Actual); Study Completion 2014-03-01 (Actual)

PRIMARY OUTCOMES:
Composite incidence of adverse device events | up to 30-days post-procedure
  The primary tolerability endpoint includes sensory nerve injury, skin necrosis, wound dehiscence, hypertrophic scarring, alopecia, surgical site infection, earlobe deformity, submental irregularity, hematomas, perforation, and palpability.

SECONDARY OUTCOMES:
Individual incidence of adverse device events | up to 3 yrs post-op
Incidence of treatment failures and cosmetic re-intervention | up to 3 yrs post-op
Quality of Life changes prior to and after surgery | up to 3 yrs post-op
Global Improvement Assessment using standardized photographic images | up to 3 yrs post-op

CONTACTS AND LOCATIONS:
Overall Officials: Martin Weisberg, MD, Study Director — Ethicon, Inc.
Locations (9):
- France (3):
  - Bernard Mole, Paris
  - Catherine Bergeret-Galley, Paris
  - Benjamin Ascher, Paris
- Germany (3):
  - Martin-Luther-Krankenhaus, Berlin
  - Chirurgie Praxisklinik Kaiserplatz, Frankfurt
  - Rotes Kreuz Krankenhous Kassel, Kassel
- Israel (2):
  - Rambam Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
- Springfield Hospital, Springfield, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not an applicable trial, product manufactured outside of US and all study sites outside US.